CLINICAL TRIAL: NCT00100074
Title: Safety and Tolerability Study of Sublingual Lobeline
Brief Title: To Assess the Safety and Tolerability of 7.5, 15 and 30 mg of Sublingual Lobeline. - 1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Purpose: Diagnostic
Other Study IDs: NIDA-CPU-0007-1
Record Dates: First submitted 2004-12-22; First posted 2004-12-23 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2004-12

CONDITIONS: Amphetamine-Related Disorders
MeSH Terms: conditions — Amphetamine-Related Disorders | interventions — Lobeline

INTERVENTIONS:
Drug: Lobeline

SUMMARY:
To assess the safety and tolerability of 7.5, 15 and 30 mg of sublingual lobeline.

DETAILED DESCRIPTION:
The primary objective of this study is to characterize the pharmacokinetics of three ascending doses of lobeline in normal volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals with a body mass index between 18 and 30.
* Willing and able to give written consent.
* Must have a negative drug test
* Females must have a negative pregnancy test prior to study drug administration
* Must have no medical contraindications as determined by routine testing

Exclusion Criteria:

* Please contact the site for more information

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8
Dates: Start 2004-09; Study Completion 2005-04

PRIMARY OUTCOMES:
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Reese Jones, M.D., Principal Investigator — Langley Porter Psychiatric Institute
Locations (1):
- U of CA, San Francisco, San Francisco, California, United States